CLINICAL TRIAL: NCT07290465
Title: Exploring Pain Perception Through Exercise-Induced Hypoalgesia Across Circadian Rhythms for Healthy Participants
Brief Title: Pain Perception and Exercise-Induced Hypoalgesia Across Circadian Rhythms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Fatema Mohamed Daoud Soliman, Principal Investigator, Medipol University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: E-10840098-202.3.02-1597
Record Dates: First submitted 2025-11-14; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Exercise Induced Hypoalgesia; Circadian Rhythm; Pain Perception; Healthy Participants; Chronotype; Physical Therapy
Keywords: Exercise-Induced Hypoalgesia; Pain Perception; Circadian Rhythm; Chronotype; Healthy Participants; High-Intensity Functional Training; Supervised Deep Breathing; Pressure Pain Threshold (PPT); Pain pressure tolerance threshold (PPTol); Quantative Sensory Testing; Bony Landmarks; Muscular Landmarks; Physical Therapy; Randomized Control Trial; Crossover; Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Participants who completed the morning sessions will cross over to the evening sessions and vice versa in a randomized order with a washout period.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both the participant and assessor will be masked to the individual's chronotype
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning Chronotype (Experimental): Participants classified as morning chronotype using the Munich Chronotype Questionnaire (MCTQ) will attend both a morning session and an evening session in randomized order with at least 72 hours between visits. Within each session the participant completes both a 12-minute supervised deep-breathing control condition and a 12-minute High-Intensity Functional Training (HIFT) intervention, separated by a 30-minute break to minimize carryover effects. Pain perception is assessed before and after each condition.
  Interventions: Behavioral: High-Intensity Functional Training (HIFT); Behavioral: Supervised Deep Breathing
- Evening Chronotype (Experimental): Participants classified as evening chronotype using the Munich Chronotype Questionnaire (MCTQ) will attend both a morning session and an evening session in randomized order with at least 72 hours between visits. Within each session the participant completes both a 12-minute supervised deep-breathing control condition and a 12-minute High-Intensity Functional Training (HIFT) intervention, separated by a 30-minute break to minimize carryover effects. Pain perception is assessed before and after each condition.
  Interventions: Behavioral: High-Intensity Functional Training (HIFT); Behavioral: Supervised Deep Breathing

INTERVENTIONS:
Behavioral: High-Intensity Functional Training (HIFT) — A 12-minute, instructor-led HIFT protocol delivered via the same video to all participants. After a 5-minute warm-up, participants perform six exercises targeting major muscle groups. The exercises are 4 lunges followed by one push-up, 10 high knees followed by 10 shuffles, burpees, squat jumps, skaters, and plank up-downs. Each exercise is done for 40 seconds then 20 seconds rest. The cycle repeats twice for a total of 12 minutes. Rate of Perceived Exertion (Borg scale) is recorded at baseline, post-warmup, during each rest interval, and immediately post-exercise. A physiotherapist supervises performance, ensures correct technique, and enforces safety and target intensity while motivating and encouraging the participant.
Behavioral: Supervised Deep Breathing — A 12-minute deep breathing session delivered via a prerecorded audio and supervised by a physiotherapist. The breathing rhythm includes inhaling for 4 seconds and exhaling for 6 seconds for a total 1 minute, followed by 1 minute of normal breathing. This cycle is repeated six times for a total duration of 12 minutes. Participants lie supine in a comfortable position and wear headphones. A self-reported Rate of Perceived Relaxation (RPR, 0-10) is recorded before and after. This serves as a non-exercise control to account for relaxation and attention effects.

SUMMARY:
The goal of this randomized crossover clinical trial is to investigate whether exercise-induced hypoalgesia (EIH) is influenced by circadian rhythm in healthy adults aged 18-40 years.

The main questions it aims to answer are:

* Does the time of day (morning vs. evening) influence changes in pain perception following exercise?
* Do chronotype, sex, or stimulation site (bony vs. muscular) alter the magnitude of this effect?

Participants will:

* Complete questionnaires
* Undergo quantitative sensory testing
* Attend both morning and evening sessions in randomized crossover order

DETAILED DESCRIPTION:
Exercise-induced hypoalgesia (EIH) is a temporary reduction in pain sensitivity following physical activity. High-intensity functional training (HIFT) has been shown to produce EIH, yet the influence of circadian rhythms on this response is not well established. Circadian timing regulates physiological processes, including pain modulation, and may contribute to variability in exercise-related analgesia.

This randomized crossover trial will examine whether time of day (morning vs. evening) affects EIH in healthy adults. It will also explore the relationship between an individual's chronotype, the efficacy of EIH and the difference in magnitude between men and women, the difference in effect between bony and muscular landmarks for pressure stimulus application.

Null Hypothesis (H0) : Circadian rhythm has no significant influence on the efficacy of exercise-induced hypoalgesia (EIH), as measured by changes in pain perception before and after high intensity functional training at different times of day (morning vs. evening).

Alternative Hypothesis (H1): Circadian rhythm significantly influences the efficacy of exercise-induced hypoalgesia (EIH), with differences in pain perception before and after high intensity functional training depending on the time of day (morning vs. evening).

Each participant will complete both morning and evening sessions in randomized order, separated by ≥72 hours. Participants who completed the morning sessions will cross over to the evening sessions and vice versa. Within each session, they will perform a 12-minute supervised deep breathing control condition and a 12-minute HIFT intervention, separated by a 30-minute rest.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* age 18 to 40 years
* good level of English that allow the enrolled participant to provide informed consent and complete the questionnaires provided
* being categorized as "moderate" in the International Physical Activity Questionnaire (IPAQ)

Exclusion Criteria:

* inability to report pain intensity reliably
* consumption of narcotics or tobacco products
* regularly taking pain medications and analgesics
* pregnant or planning to get pregnant
* surgery within the last 12 months
* acute or chronic pain conditions
* uncontrolled hypertension
* cardiovascular diseases, pulmonary diseases, neurological diseases with significant changes in somatosensory and pain perception, metabolic diseases, serious systemic diseases or conditions that restrict normal daily activities, inflammatory conditions (e.g. rheumatoid arthritis), or orthopedic injuries
* intolerable pain during the pain perception test
* serious psychiatric conditions (e.g., schizophrenia and bipolar disorder) or psychological disorders (e.g., depression) that may affect pain thresholds (16).
* Severe sleep disorders and circadian rhythm disturbances
* BMI > 30
* serious fatigue or delayed-onset muscle soreness (9) at least 24 h after exercise sessions or a sudden change in activity for more than one week

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Threshold (PPT) | Baseline (0 minute before intervention) and immediately post-intervention (within 2 minutes) Measured in both high intensity functional training (HIFT) and supervised deep-breathing conditions during each morning and evening session
  Pressure Pain Threshold (PPT) will be measured using an algometer at standardized bony and muscular landmarks. Pressure Pain Threshold (PPT) is defined as the minimal pressure at which a participant first perceives pain. Changes in Pressure Pain Threshold (PPT) will be used to assess the magnitude of exercise-induced hypoalgesia (EIH).
  Unit: kg/cm²
Pressure Pain Tolerance (PPTol) | Baseline (0 minute before intervention) and immediately post-intervention (within 2 minutes) Measured in both high intensity functional training (HIFT) and supervised deep-breathing conditions during each morning and evening session
  Pressure Pain Tolerance (PPTol) will be measured using an algometer at standardized bony and muscular landmarks. Pressure Pain Tolerance (PPTol) is defined as the maximal pressure the participant is willing to tolerate. Changes in Pressure Pain Tolerance (PPTol) will be used to assess pain modulation in response to exercise across circadian phases.
  Unit: kg/cm²

SECONDARY OUTCOMES:
Munich Chronotype Questionnaire (MCTQ) | Baseline (before any intervention session)
  Chronotype will be assessed using the Munich Chronotype Questionnaire (MCTQ). Participants will be classified as morning or evening chronotypes to examine whether individual circadian preference moderates exercise-induced hypoalgesia.
Pain Catastrophizing (PCS) | Baseline (before any intervention session)
  Pain-related cognitions will be measured using the Pain Catastrophizing Scale (PCS) to control for potential psychological influences and understandings on pain perception. PCS is scored according to a 5-point Likert scale ranging from 0 = not at all to 4 = all the time with a maximum score of 52, with higher scores >30 indicating increased pain catastrophizing.
Fear of Pain (FPQ-9) | Baseline (before any intervention session)
  Fear of pain will be assessed using the Fear of Pain Questionnaire-9 (FPQ-9), as psychological fear responses may influence pain reporting. Fear of Pain Questionnaire-9 (FPQ-9) is scored by using a 5-point Likert scale with a score ranging from 9 to 45 with higher scores indicate greater fear of pain.
Brief Version of the Pittsburgh Sleep Quality Index (B-PSQI) | Baseline (before any intervention session)
  The Brief Pittsburgh Sleep Quality Index (B-PSQI) will be used to assess participants' sleep patterns and their potential influence on pain modulation. Total score ranges between 0 and 15, where higher values suggest worse quality of sleep. Scores from 0 to 5 indicate good sleep quality and scores of ≥6 poor sleep quality.
Depression Anxiety Stress Scales (DASS-21) | Baseline (before any intervention session)
  Depression, Anxiety, and Stress Scale-21 (DASS-21) will be administered to capture psychological states that may influence experimental pain measures. Scores are presented as a total score (between 0 and 63) and a score for the three subscales (between 0 and 21). Higher scores indicate worse psychological distress.
Rate of Perceived Exertion (RPE, Borg scale) | At minute 0 (before warm-up), at minute 5 (after warm-up), every 1 minute during the high-intensity functional training (HIFT) protocol, and at minute 17 (end of session).
  Rate of Perceived Exertion (RPE, Borg scale) will be recorded during High intensity functional training (HIFT) to confirm intensity differences between interventions. A scale of 0-10 (1 being very light, and 10 being maximum effort) is used.
Rate of Perceived Relaxation (RPR) | At minute 0 (baseline) and at minute 12 (immediately after the supervised deep-breathing session).
  Relaxation level during supervised deep breathing control session will be assessed using a 0-10 relaxation scale. The score range is 0 (no relaxation) to 10 (maximum relaxation) with higher scores indicate better relaxation.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Ergezen Şahin, Dr. Assistant Professor, Study Director — Department of Physiotherapy and Rehabilitation/Istanbul Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The revised International Association for the Study of Pain definition of pain: concepts, challenges, and compromises. — https://doi.org/10.1097/j.pain.0000000000001939
- See also: A meta-analytic review of the hypoalgesic effects of exercise — https://doi.org/10.1016/j.jpain.2012.09.006
- See also: Exercise induced hypoalgesia after a high intensity functional training: a randomized controlled crossover study — https://doi.org/10.1186/s13102-024-00969-4
- See also: Quantitative sensory testing: a practical guide and clinical applications — https://doi.org/10.1016/j.bjae.2024.05.004
- See also: Day-to-day reliability of pressure pain threshold and pain ratings in college-aged men. International journal of rehabilitation research. — https://doi.org/10.1097/MRR.0000000000000111
- See also: New Insights Into the Circadian Rhythm and Its Related Diseases. — https://doi.org/10.3389/fphys.2019.00682